CLINICAL TRIAL: NCT01679249
Title: Blood Volume Analysis and Related Outcomes in Hemodialysis
Status: Completed | Type: Observational
Sponsor: VA New York Harbor Healthcare System (U.S. Federal Agency)
Collaborators: Daxor Corporation (Industry)
Responsible Party: Principal Investigator, David S. Goldfarb, M.D., Chief, Nephrology, VA New York Harbor Healthcare System
Other Study IDs: 01249
Record Dates: First submitted 2012-08-31; First posted 2012-09-05 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: End Stage Kidney Disease
Keywords: extracellular fluid volume; hypotension; hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Hypotension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hemodialysis patients: Stable prevalent patients on 3-times-per-week hemodialysis

SUMMARY:
An understanding of fluid changes that occur during hemodialysis (HD) with ultrafiltration (UF) is essential for determining the efficacy of HD, as well as for reducing complications related to hypovolemia or, conversely, chronic volume overload.

DETAILED DESCRIPTION:
Background: Accurate assessment of the BV and distribution of body fluids is essential for prescribing HD and for reducing complications related to hypovolemia and volume overload. Monitoring relative changes in BV using hematocrit (Hct), e.g. CLM-III, an indirect method, cannot be used to determine the absolute levels of BV. Here we report the first study of isotope BV measurement (IBVM) for assessing volume status in HD patients using indicator dilutional method.

10 adult HD patients were enrolled in this prospective observational study. Multi-point IBVM before and after HD was performed using BVA-100 (Daxor, New York, NY). BVA-100 calculates BV with an accuracy of ±2.5%, by using <25μCi of iodinated I-131 albumin. It assumes normal BV for a given individual on the basis of patients' deviation from ideal body weight. Fluid loss from the extravascular component of the extracellular space (EV) was calculated by subtracting absolute BV change from total weight loss. Intradialytic relative BV changes were measured by CLM-III during the same HD session. Bland-Altman plot was used to compare relative BV change pre- and post-HD by IBVM and CLM-III.

ELIGIBILITY:
Inclusion Criteria:

* Age >21 years
* Primary diagnosis of either chronic or acute kidney disease
* Currently receiving HD treatment
* Thrice-weekly or twice-weekly HD schedule
* Treated with standard bicarbonate HD for at least the preceding 6 months

Exclusion Criteria:

* Pregnant women or nursing mothers
* Known hypersensitivity to iodine, eggs, albumin or any other component of the Volumex injection kit
* Current enrollment in another investigational treatment protocol for dialysis
* The need to perform hemodialysis with predilution because this will interfere with measurements of relative blood volume changes (ΔRBV)
* Kidney transplantation
* Malignancy requiring chemotherapy
* Unmeasurable blood pressure with a sphygmomanometer
* Active hematological disease
* Active gastrointestinal bleeding
* Severe malnutrition (predialysis serum albumin <2.6 g/dL)
* Persistent condition of intradialytic blood pressure instability (hypotensive episodes in >80% of regular dialysis sessions) within the previous one month period

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the pool of patients at the Dialysis Center at the Department of Veteran Affairs New York Harbor Healthcare System who are currently undergoing dialysis for treatment of chronic kidney disease.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Blood volume measurement and comparison to Crit-Line reading | Six months
  To compare the results obtained by two different methods of assessing BV: direct measurement of BV using the Blood Volume Analyzer (BVA-100) vs. indirect measurement of relative changes in BV using the Crit-Line Monitor (CLM III). Blood volume is measured in liters and compared with "ideal blood volume" nomograms. Crit-Line Monitor measures relative change in blood volume as a percentage change and does not have absolute values.

CONTACTS AND LOCATIONS:
Overall Officials: David S Goldfarb, MD, Principal Investigator — VA New York Harbor Healthcare System
Locations (1):
- New York Harbor VA Healthcare System Hemodialysis Unit, New York, New York, United States